CLINICAL TRIAL: NCT05644587
Title: Novel Induction to Buprenorphine/Naloxone: A Quasi-Experimental Study With Comparison Group
Brief Title: Novel Induction to Buprenorphine/Naloxone
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment numbers
Sponsor: Bicycle Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bicycle-005
Record Dates: First submitted 2022-11-21; First posted 2022-12-09 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Opioid Use Disorder; Opioid Use; Opioid Abuse; Opioid Misuse; Opioid Dependence
Keywords: opioid; opioid use disorder; buprenorphine; microdosing
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Induction Arm (Active Comparator): In this arm, study participants will wait until they have significant opioid withdrawal (SOWS score >=17) prior to starting buprenorphine. Participants will then started with 2 mg sublingual and escalate to a maximum of 12 mg on the first day depending on withdrawal symptoms. On day 2, the participant will take same dose as the total dose taken on day 1, and continue that dose daily until reevaluation.
  Interventions: Drug: buprenorphine/naloxone
- Microdosing Induction Arm (Active Comparator): In this arm, study participants will not wait until they have significant opioid withdrawal. They will take 0.5 mg buprenorphine on day 1, 2 mg on day 2, 4 mg on day 3, 6 mg on day 4, 8 mg on day 5 and 12 mg starting on day 6.
  Interventions: Drug: buprenorphine/naloxone

INTERVENTIONS:
Drug: buprenorphine/naloxone — Buprenorphine/naloxone will be used to begin each patient's treatment for opioid use disorder.

SUMMARY:
Microdosing induction is a novel method of starting buprenorphine/naloxone without patients experiencing the opioid withdrawal that is a part of traditional induction. Patients take small doses of buprenorphine/naloxone that increase slowly over a week. Although microdosing induction has been supported anecdotally, its effectiveness is not known. The proposed study will compare the effectiveness and safety of two induction strategies for transitioning patients from opioids to buprenorphine/naloxone. All inductions will occur in an outpatient telehealth opioid use disorder (OUD) treatment setting. The study will compare patients who receive traditional induction versus microdosing induction. Primary outcomes include effectiveness and safety. Secondary outcomes include treatment retention, self-reported use of opioids during induction, return to opioid use, opioid appearance in drug screens, craving/withdrawal symptoms, and patient satisfaction.

DETAILED DESCRIPTION:
Medication for OUD (MOUD) is a first-line treatment for OUD and improves outcomes in mortality, retention in treatment, and non-prescribed opioid use. Buprenorphine/naloxone is the only MOUD of the three FDA-approved medications for OUD available in the telehealth setting, as methadone and injectable naltrexone must be managed in an in-person setting. Buprenorphine/naloxone, also referred to as brand name Suboxone, is administered by placing a film strip under the tongue. Buprenorphine acts as a partial agonist with a high binding affinity at the mu-opioid receptor; clearance of the pure opioid agonist must occur before a full dose of buprenorphine is administered, as buprenorphine will displace opioid agonists with lower binding affinity at the receptor and cause rapid-onset "precipitated withdrawal." During traditional induction, patients must abstain from opioids prior to starting buprenorphine/naloxone and thus endure mild-to-moderate opioid withdrawal before initiating buprenorphine (to avoid precipitated withdrawal). Barriers to traditional induction include the required withdrawal period, fear of precipitated withdrawal (particularly with increased fentanyl in the opioid supply, which is lipophilic and thus remains in the body longer after last use), and an intolerable withdrawal period (which increases the risk of a patient leaving treatment to return to non-prescribed opioid use). In addition, there are patients who are not ready to stop their opioid but are ready to start treatment.

First described in the literature as the Bernese Method in 2016, microdosing induction was developed to overcome these barriers. Microdosing induction requires the administration of small but escalating doses of buprenorphine/naloxone over a period of several days to weeks, such that the buprenorphine slowly overcomes the effect of the opioid agonist at the receptor. This technique does not require a period of withdrawal prior to starting treatment. Various microdosing induction protocols have been described primarily in inpatient settings in case reports, case series, and literature reviews. No published research studies exist that systematically evaluate the effectiveness and safety of microdosing induction, particularly in a telehealth setting.

Using a quasi-experimental design for evaluating MOUD induction strategies in a telehealth setting, the investigators will estimate the effect of microdosing induction on patient completion of successful induction with mild withdrawal, adjusted maximum withdrawal score, and adverse events. The investigators hypothesize that microdosing induction patients will have higher odds of completing a successful induction with mild withdrawal, lower maximum withdrawal scores, and a similar number of adverse events compared to traditional induction patients.

Study Details:

The proposed study will follow a quasi-experimental design with a comparison group to evaluate the effectiveness and safety of microdosing induction versus traditional induction of buprenorphine/naloxone in telehealth patients at Bicycle Health. Bicycle Health is a digital health company that provides biopsychosocial treatment of OUD via telehealth. With guidance from the research team, participating medical providers at Bicycle Health will recruit patients at intake who meet eligibility criteria (see Participant Population section below). Based on sample size calculations under different scenarios, and feasibility given current intake rates at Bicycle Health, the study will enroll at least 85 patients in the microdosing induction group, and at least 85 patients in the comparison group.

The study period will take place during the induction period of treatment. All enrolled patients will undergo assessment by a participating provider through a visit at days one, four, seven, and ten, which will include a modified-clinical opiate withdrawal scale (M-COWS) and a clinical interview. Day one for microdosing induction patients will be the first day they begin taking buprenorphine/naloxone. Day one for the traditional induction study arm will be the first day without opioids. Surveys will be completed by the providers during each visit. The patient will also undergo daily self-assessments for 10 days, which will include subjective opiate withdrawal scale (SOWS), presence of cravings, self-reported continued opioid use, and patient satisfaction.

After the induction period, two urine drug screens will be conducted to monitor opioid use in early treatment. Patients at Bicycle Health receive four urine drug screen cups and four fentanyl dip cards in the mail about 1 week after their first appointment. The first urine drug screen is expected to be completed when it is delivered to the patient's residence, and it will primarily be used to ensure patients are taking buprenorphine. The second urine drug screen is expected to be completed between 14-21 days after the first test is completed. This urine drug screening will be used to collect objective data on opioid use after initiation of buprenorphine. Retention in treatment will be measured at day 10 and day 30.

Primary outcomes assess effectiveness and safety:

* Completion of induction with no/mild withdrawal: receiving ≥ 8 mg of buprenorphine/naloxone with no concurrent self-reported use of opioids by the end of induction and M-COWS score remains in mild withdrawal range defined as ≤ 12 points throughout induction
* Maximum M-COWS score minus baseline M-COWS
* Average and median M-COWS scores at day 1,4,7,10
* Average and median SOWS scores ≤12 daily
* All adverse events, defined as:
* An untoward medical occurrence as a study participant that was administered a study intervention, which does not necessarily have a causal relationship with this intervention
* An untoward medical occurrence meeting one of the following criteria at any dose - results in death, is life-threatening, requires inpatient hospitalization, results in persistent or significant disability or incapacity

Secondary outcomes include:

* Treatment retention: defined as patient attendance at visit with a participating provider on day 10 (+5) and day 30 (+7)
* Self-reported return to opioid use after induction
* Opioid appearance in drug screens
* Self-reported cravings
* Patient satisfaction

The investigators will use a multilevel logistic regression model to estimate the odds of completing a successful induction with mild withdrawal. The investigators will use a multilevel cox proportional hazards regression model for retention analysis. All models will adjust for covariates. Covariates may include age, sex, payment method, baseline M-COWS score. Additional covariates collected through patient intake form will be considered, including history of unsuccessful induction, history of precipitated withdrawal, and history of experience with buprenorphine. A difference-in-difference analysis using multilevel linear regression will be used to assess maximum M-COWS score minus baseline M-COWS score. Covariates will be adjusted for in the model. Covariates may include age, sex, payment method, baseline M-COWS score, history of unsuccessful induction, history of precipitated withdrawal, and history of experience with buprenorphine. Average and median M-COWS and SOWS will be calculated at each data collection timepoint. Adverse events will be reported as a percentage of enrolled patients who experienced an adverse event. For secondary outcomes, level of craving/withdrawal symptoms and patient satisfaction, the investigators will calculate the mean and median scores for outcomes at each measurement time point.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment with Bicycle Health services
* Aged 18 years old or older
* Diagnosis of opioid use disorder confirmed by DSM-5 criteria
* In no/mild withdrawal at the time of intake
* Need to undergo induction to buprenorphine from a full opioid agonist
* Use of full opioid agonists not directly from a pharmacy within the last 24 hours
* Pharmacy stock check of 2 mg film/tablet done before visit
* Willingness and ability to follow study protocols, and the ability to provide informed consent

Exclusion Criteria:

* Known allergy or sensitivity to buprenorphine/naloxone
* Any circumstance that precludes the need for induction
* In moderate to severe withdrawal at the time of intake
* Severe or complex medical/psychiatric comorbidity that requires a customized induction schedule or surveillance
* Any element that would exclude an individual from Bicycle Health services in general (e.g., homelessness, severe untreated mental illness)
* Patients requesting specific induction technique
* Patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete induction with no/mild withdrawal | 10 days
  Completion of induction with no/mild withdrawal
Modified-Clinical Opiate Withdrawal Scale (M-COWS) scores | 10 days
  Average/median and Maximum M-COWS scores for each participant. Scores range from 0-48, with higher scores indicating more withdrawal symptoms.
Subjective Opiate Withdrawal Scale (SOWS) scores | 10 days
  Average/median SOWS scores for each participant. Score range from 0-64, with higher scores indicating more withdrawal symptoms.
Adverse outcomes | 10 days
  Any untoward medial occurrence

SECONDARY OUTCOMES:
Treatment retention | 30 days
  Patient attendance at visit with a participating provider on day 10 and day 30
Opioid use | 30 days
  Self-reported return to opioid use after buprenorphine/naloxone induction
Toxicology screens | 30 days
  Opioid appearance in drug screens
Cravings | 30 days
  Patient self-reported opioid-related cravings
Patient satisfaction | 30 days
  On a scale of 1 (highly unsatisfactory) to 5 (highly satisfactory), participants will be asked to rate their satisfaction with the buprenorphine induction process.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Weiner, MD, MPH, Principal Investigator — Bicycle Health
Locations (1):
- Bicycle Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammig R, Kemter A, Strasser J, von Bardeleben U, Gugger B, Walter M, Dursteler KM, Vogel M. Use of microdoses for induction of buprenorphine treatment with overlapping full opioid agonist use: the Bernese method. Subst Abuse Rehabil. 2016 Jul 20;7:99-105. doi: 10.2147/SAR.S109919. eCollection 2016. PMID 27499655
- See also: Related Info — https://www.bicyclehealth.com/research